CLINICAL TRIAL: NCT02902965
Title: An Open-label Study of Ibrutinib in Combination With Bortezomib and Dexamethasone in Subjects With Relapsed or Relapsed and Refractory Multiple Myeloma
Brief Title: Study of Ibrutinib in Combination With Bortezomib and Dexamethasone in Subjects With Relapsed/Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics Switzerland GmbH (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1139-CA
Record Dates: First submitted 2016-08-19; First posted 2016-09-16 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma
Keywords: Bruton's Tyrosine Kinase; Bortezomib; Dexamethasone; Ibrutinib
MeSH Terms: conditions — Multiple Myeloma | interventions — ibrutinib; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib+ Bortezomib+ Dexamethasone (Experimental)
  Interventions: Drug: Ibrutinib; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib 840 mg orally, once daily continuously starting day 1 of cycle 1 until confirmed disease progression, unacceptable toxicity or other protocol specified reason for discontinuation
  Other Names: Imbruvica
Drug: Bortezomib — Cycles 1-8: (21-day cycle): Bortezomib 1.3 mg/m^2 sub-cutaneously on days 1, 4, 8, and 11 of each Cycle Cycles 9-12: (42-day cycle): Bortezomib 1.3 mg/m^2 sub-cutaneously on days 1, 8, 22 and 29 of each Cycle
  Other Names: Velcade
Drug: Dexamethasone — Cycles 1-8: (21-day cycle): Dexamethasone 20 mg orally on days 1, 2, 4, 5, 8, 9, 11 and 12 of each cycle Cycles 9-12: (42-day cycle): Dexamethasone 20 mg orally on days 1, 2, 8, 9, 22, 23, 29 and 30 of each cycle Cycles 13+ (28-day cycle): Dexamethasone 40 mg orally once weekly
  Dose adjustment of dexamethasone to 10 mg on days specified during cycles 1-12 and 20 mg weekly during cycles 13+ is recommended for subjects >75 years of age.
  Following implementation of Protocol Amendment 4, dexamethasone administration was reduced to Days 1, 4, 8 and 11 during each 21-day cycle (Cycles 1-8) and on Days 1, 8, 22, 29 on each 42-day cycle (Cycles 9-12) and unchanged thereafter.

SUMMARY:
This is a Phase 2 open-label study to evaluate the efficacy and safety of ibrutinib in combination with bortezomib and dexamethasone for patients with relapsed or relapsed and refractory multiple myeloma.

DETAILED DESCRIPTION:
Bruton's tyrosine kinase (Btk) is an enzyme that is present in hematopoeitic cells other than T cells and is necessary for downstream signal transduction from various hematopoietic receptors including the B cell receptor as well as some Fc, chemokine and adhesion receptors, and is crucial for both B cell development and osteoclastogenesis. Although down-regulated in normal plasma cells, Btk is highly expressed in the malignant cells from many myeloma patients and some cell lines. Ibrutinib is a potent and specific inhibitor of Btk currently in Phase 2 and 3 clinical trials. The current study is designed and intended to determine the safety and efficacy of ibrutinib in combination with bortezomib and dexamethasone in subjects with relapsed/relapsed and refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with multiple myeloma (MM) who have received 1-3 prior lines of therapy and have demonstrated disease progression since the completion of the most recent treatment regimen. (Subjects may have received prior bortezomib exposure if it does not meet the exclusion criteria for prior proteasome inhibitor use)
* Measurable disease defined by at least one of the following:

  * Serum monoclonal protein (SPEP) ≥1 g/dL (for subjects with immunoglobulin A (IgA), immunoglobulin D (IgD), immunoglobulin E (IgE) or immunoglobulin M (IgM) multiple myeloma SPEP ≥0.5 g/dL)
  * Urine monoclonal protein (UPEP) ≥200 mg by 24 hour urine electrophoresis
* Adequate hematologic, hepatic and renal function
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2

Exclusion Criteria:

* Subject must not have primary refractory disease
* Refractory or non-responsive to prior proteasome inhibitor (PI) therapy (bortezomib or carfilzomib)
* Peripheral neuropathy Grade ≥2 or Grade 1 with pain at Screening
* Plasma cell leukemia, primary amyloidosis, or POEMS syndrome
* Unable to swallow capsules or disease significantly affecting gastrointestinal function
* Requires treatment with strong CYP3A inhibitors
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Hauns, MD, Study Director — Pharmacyclics Switzerland GmbH
Locations (33):
- Czechia (4):
  - Fakultní nemocnice Brno, Brno
  - Fakultní nemocnice Hradec Králové, Nový Hradec Králové
  - Fakultní nemocnice Ostrava, Ostrava-Poruba
  - Všeobecná fakultní nemocnice v Praha, Prague
- Germany (4):
  - Helios-Kliniken Berlin-Buch, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Universitätsklinikum Jena, Jena
  - Klinikum der Universität München Campus Grosshadern, München
- Greece (6):
  - 251 General Air Force Hospital, Athens
  - General Hospital of Athens "Alexandra", Athens
  - General Hospital of Athens "Evangelismos", Athens
  - General Hospital of Athens "LAIKO", Athens
  - University General Hospital of Patra, Pátrai
  - General Hospital of Thessaloniki "G. Papanikolau", Thessaloniki
- Italy (6):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Istituto Scientifico Romagnolo Per lo Studio e la Cura dei Tumori, Meldola (FC)
  - Ospedale Santa Maria delle Croci, Ravenna
  - Ospedale degli Infermi, Rimini
  - Azienda Ospedaliera S. Maria di Terni, Terni
- Spain (9):
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - ICO Badalona-Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Dr. Peset, Valencia
- Turkey (Türkiye) (4):
  - Ankara University Medical Faculty, Ankara
  - Dokuz Eylul University Medicine Faculty, Izmir
  - Erciyes University Medical Faculty, Kayseri
  - Ondokuz Mayis Univ. Med. Fac., Samsun

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib+ Bortezomib+ Dexamethasone: Ibrutinib (I): I 840 mg orally, once daily continuously starting day 1 of Cycle (C) 1 until confirmed disease progression, unacceptable toxicity or other protocol specified reason for discontinuation Bortezomib (B): C 1-8: (21-day C): B 1.3 mg/m^2 sub-cutaneously on days 1, 4, 8, and 11 of each C C 9-12: (42-day C): B 1.3 mg/m^2 sub-cutaneously on days 1, 8, 22 and 29 of each C Dexamethasone (D): C 1-8: (21-day C): D 20 mg orally on days 1, 2, 4, 5, 8, 9, 11 and 12 of each C C 9-12: (42-day C): D 20 mg orally on days 1, 2, 8, 9, 22, 23, 29 and 30 of each C C 13+ (28-day C): D 40 mg orally once weekly Dose adjustment of D to 10 mg on days specified during C 1-12 and 20 mg weekly during C 13+ is recommended for subjects >75 years of age.
  Following implementation of Protocol Amendment4, D administration was reduced to Days 1, 4, 8, and 11 during each 21-day C (C 1-8) and on Days 1, 8, 22 and 29 on each 42-day C (C 9-12) and unchanged thereafter
Period: Overall Study
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
Started | 74
Completed | 64
Not Completed | 10
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Population: All participant received: see description on Arm/Group description.
Groups:
- Ibrutinib+ Bortezomib+ Dexamethasone: Ibrutinib (I): I 840 mg orally, once daily continuously starting day 1 of Cycle (C) 1 until confirmed disease progression, unacceptable toxicity or other protocol specified reason for discontinuation Bortezomib (B): C 1-8: (21-day C): B 1.3 mg/m^2 sub-cutaneously on days 1, 4, 8, and 11 of each C C 9-12: (42-day C): B 1.3 mg/m^2 sub-cutaneously on days 1, 8, 22 and 29 of each C Dexamethasone(D): C 1-8: (21-day C): D 20 mg orally on days 1, 2, 4, 5, 8, 9, 11 and 12 of each C C 9-12: (42-day C): D 20 mg orally on days 1, 2, 8, 9, 22, 23, 29 and 30 of each C C 13+ (28-day C): D 40 mg orally once weekly Dose adjustment of D to 10 mg on days specified during C 1-12 and 20 mg weekly during C 13+ is recommended for subjects >75 years of age.
  Following implementation of Protocol Amendment 4, D administration was reduced to Days 1, 4, 8 and 11 during each 21-day C (C 1-8) and on Days 1, 8, 22 and 29 on each 42-day C (C 9-12) and unchanged thereafter.
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 71
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Greece | 11
  Turkey | 13
  Czechia | 23
  Italy | 10
  Germany | 1
  Spain | 16

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival (PFS)
Description: The primary efficacy endpoint of this study is mPFS. Progression free survival is defined as the time from the date of first dose of study treatment to confirmed disease progression or death from any cause, whichever occurs first.
Time Frame: The median time on study was 19.6 months (range: 0.16+, 24.64). Participants were evaluated for Progression-Free Survival (PFS) during their entire time on the study.
Population: All participant received: see description on Arm/Group description. Following implementation of Amendment 4, dexamethasone administration was reduced to Days 1, 4, 8 and 11 during each 21-day cycle (Cycles 1-8) and on Days 1, 8, 22 and 29 on each 42-day cycle (Cycles 9-12) and unchanged thereafter.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ibrutinib+ Bortezomib+ Dexamethasone: Ibrutinib (I): I 840 mg orally, once daily continuously starting day 1 of Cycle (C) 1 until confirmed disease progression, unacceptable toxicity or other protocol specified reason for discontinuation Bortezomib (B): C 1-8: (21-day C): B 1.3 mg/m^2 sub-cutaneously on days 1, 4, 8, and 11 of each C C 9-12: (42-day C): B 1.3 mg/m^2 sub-cutaneously on days 1, 8, 22 and 29 of each C Dexamethasone (D): C 1-8: (21-day C): D 20 mg orally on days 1, 2, 4, 5, 8, 9, 11 and 12 of each C C 9-12: (42-day C): D 20 mg orally on days 1, 2, 8, 9, 22, 23, 29 and 30 of each C C 13+ (28-day C): D 40 mg orally once weekly Dose adjustment of D to 10 mg on days specified during C 1-12 and 20 mg weekly during C 13+ is recommended for subjects >75 years of age.
  Following implementation of Protocol Amendment 4, D administration was reduced to Days 1, 4, 8, and 11 during each 21-day C (C 1-8) and on Days 1, 8, 22 and 29 on each 42-day C (C 9-12) and unchanged thereafter
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
Number analyzed (Participants) | 74
Months | 8.5 [6.2 to 10.8]
Statistical Analysis 1: Comparison: Ibrutinib+ Bortezomib+ Dexamethasone; Test type: Other; median PFS = 8.5, 95% CI 2-sided [6.2 to 10.8] — Kaplan-Meier estimates for median PFS and its associated 95% confidence intervals using log-log transformed Greenwood variance estimate were calculated

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate is the percentage of participants who achieve a PR or better over the course of the study but prior to initiation of subsequent anti-cancer therapy
Time Frame: The median time on study was 19.6 months (range: 0.16+, 24.64). Participants were evaluated for Overall Response (OR) during the entire time on the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
Number analyzed (Participants) | 74
percentage of participants | 56.8 [44.7 to 68.2]
Statistical Analysis 1: Comparison: Ibrutinib+ Bortezomib+ Dexamethasone; Test type: Other; ORR in % = 56.8, 95% CI 2-sided [44.7 to 68.2] — Overall response = confirmed sCR + CR + VGPR + PR with corresponding 95% Exact binomial Cl

3. Secondary Outcome: Progression Free Survival (PFS) at Landmark Points - 20 Months
Description: PFS at landmark points are the percentage of participants without progression (i.e., KM estimates) at the landmark time endpoints.
Time Frame: The median time on study was 19.6 months (range: 0.16+, 24.64), with the 20 month Progression-Free Survival (PFS) rate presented based on Kaplan-Meier estimates.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
Number analyzed (Participants) | 74
percentage of participants | 6.6 [1.6 to 16.9]
Statistical Analysis 1: Comparison: Ibrutinib+ Bortezomib+ Dexamethasone; Test type: Other; PFS rate = 6.6, 95% CI 2-sided [1.6 to 16.9] — Kaplan-Meier method used for PFS rate and its associated 95% confidence intervals using log-log transformed Greenwood variance estimate were calculated

4. Secondary Outcome: Duration of Response (DOR)
Description: The time interval between the date of initial documentation of a response (PR or better) and the date of first documented evidence of PD, death, or date of censoring for the participants not progressed/died. The censoring date is the last adequate tumor assessment date.
Time Frame: The median time on study was 19.6 months (range: 0.16+, 24.64).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
Number analyzed (Participants) | 74
Months | 9.5 [6.9 to 10.6]

5. Secondary Outcome: Overall Survival (OS) at 24 Months
Description: As the median overall survival has not been reached, the data for the landmark analysis at 24 months are provided.
Time Frame: The median time on study was 19.6 months (0.16+, 24.64), with the 24 month Overall Survival (OS) rate presented based on Kaplan-Meier estimates.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
Number analyzed (Participants) | 74
percentage of participants | 53.6 [38.0 to 67.0]

6. Secondary Outcome: Time to Progression (TTP)
Description: Time from date of first dose of study treatment to the date of first documented evidence of PD or date of censoring for the participants not progressed. The censoring date is the last adequate tumor assessment date.
Time Frame: The median time on study was 19.6 months (range: 0.16+, 24.64).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
Number analyzed (Participants) | 74
Months | 10.6 [7.8 to 12]
Statistical Analysis 1: Comparison: Ibrutinib+ Bortezomib+ Dexamethasone; Test type: Other; median TTP = 10.6, 95% CI 2-sided [7.8 to 12] — KM estimates for median TTP with associated 95% CI

7. Secondary Outcome: Safety and Tolerability of Ibrutinib in Combination With Bortezomib and Dexamethasone as Measured by the Number of Participants With Adverse Events.
Description: Safety and tolerability of ibrutinib in combination with bortezomib and dexamethasone as measured by the frequency and type of adverse events graded using the NCI CTCAE v 4.03. Frequency and Type of Adverse Events are reported in the Adverse Events module
Time Frame: From first dose of Ibrutinib to within 30 days of last dose for each participant or until study closure. This is the median treatment duration for Ibrutinib of 5.7 months (range: 0.1 - 23.7 months) +30 days (Adverse Events collection period).
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Ibrutinib+ Bortezomib+ Dexamethasone: Ibrutinib (I): I 840 mg orally, once daily continuously starting day 1 of Cycle (C) 1 until confirmed disease progression, unacceptable toxicity or other protocol specified reason for discontinuation Bortezomib (B): C 1-8: (21-day C): B 1.3 mg/m^2 sub-cutaneously on days 1, 4, 8, and 11 of each C C 9-12: (42-day C): B 1.3 mg/m^2 sub-cutaneously on days 1, 8, 22 and 29 of each C Dexamethasone (D): C 1-8: (21-day C): D 20 mg orally on days 1, 2, 4, 5, 8, 9, 11 and 12 of each C C 9-12: (42-day C): D 20 mg orally on days 1, 2, 8, 9, 22, 23, 29 and 30 of each C C 13+ (28-day C): D 40 mg orally once weekly Dose adjustment of D to 10 mg on days specified during C 1-12 and 20 mg weekly during C 13+ is recommended for subjects >75 years of age.
  Following implementation of Protocol Amendment 4, D administration was reduced to Days 1, 4, 8 and 11 during each 21-day C (C 1-8) and on Days 1, 8, 22 and 29 on each 42-day C (C 9-12) and unchanged thereafter.
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
Number analyzed (Participants) | 74
Participants | 74

ADVERSE EVENTS:
Time Frame: From first dose of Ibrutinib to within 30 days of last dose for each participant or until study closure. This is the median treatment duration for Ibrutinib of 5.7 months (range: 0.1 - 23.7 months) +30 days (Adverse Events collection period).
Description: Number of participants who had experienced at least one treatment emergent AE.
Arm/Group | Ibrutinib+ Bortezomib+ Dexamethasone
All-Cause Mortality (participants affected / at risk) | 27/74
Serious Adverse Events (participants affected / at risk) | 47/74
Other Adverse Events (participants affected / at risk) | 74/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib+ Bortezomib+ Dexamethasone (N=74)
Circulatory collapse (Vascular disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Decrease appetite (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Bronchitis viral (Infections and infestations) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Haemophilus bacteraemia (Infections and infestations) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Pneumococcal sepsis (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 11 (12)
Pneumonia bacterial (Infections and infestations) | 2 (2)
Pneumonia escherichia (Infections and infestations) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 2 (2)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (4)
Staphylococcal infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Spontaneous haematoma (Blood and lymphatic system disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib+ Bortezomib+ Dexamethasone (N=74)
Hypertension (Vascular disorders) | 10 (14)
Hypotension (Vascular disorders) | 8 (9)
Asthenia (General disorders) | 22 (60)
Fatigue (General disorders) | 21 (40)
Oedema peripheral (General disorders) | 21 (29)
Pain (General disorders) | 3 (3)
Peripheral swelling (General disorders) | 5 (6)
Pyrexia (General disorders) | 13 (18)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6)
Blood creatinine increased (Investigations) | 4 (6)
Weight decreased (Investigations) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 28 (66)
Lymphopenia (Blood and lymphatic system disorders) | 11 (50)
Neutropenia (Blood and lymphatic system disorders) | 10 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 45 (293)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 6 (6)
Neuropathy peripheral (Nervous system disorders) | 4 (6)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 5 (14)
Periperal sensory neuropathy (Nervous system disorders) | 18 (19)
Polyneuropathy (Nervous system disorders) | 5 (10)
Somnolence (Nervous system disorders) | 4 (6)
Syncope (Nervous system disorders) | 4 (4)
Lacrimation increased (Eye disorders) | 4 (5)
Vision blurred (Eye disorders) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (8)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 10 (17)
Diarrhoea (Gastrointestinal disorders) | 40 (119)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Mouth haemorrhage (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 18 (24)
Stomatitis (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 11 (13)
Renal impairment (Renal and urinary disorders) | 3 (6)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (22)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (19)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8)
Cushingoid (Endocrine disorders) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 10 (11)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (22)
Hypocalcaemia (Metabolism and nutrition disorders) | 11 (16)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (10)
Platelet count decreased (Investigations) | 4 (16)
Bronchitis (Infections and infestations) | 9 (11)
Conjunctivitis (Infections and infestations) | 10 (11)
Herpes zoster (Infections and infestations) | 3 (4)
Infection (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 10 (17)
Oral candidiasis (Infections and infestations) | 4 (4)
Pharyngitis (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 5 (5)
Respiratory tract infection (Infections and infestations) | 7 (11)
Tonsillitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 19 (29)
Urinary tract infection (Infections and infestations) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT02902965/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT02902965/SAP_001.pdf